CLINICAL TRIAL: NCT06353282
Title: 3, 4-methylenedioxymethamphetamine (MDMA) for Treatment-resistant Post-traumatic Stress Disorder (PTSD) in Adolescents
Brief Title: MDMA-Assisted Psychotherapy for Treatment Resistant PTSD in Adolescents
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Under review with FDA
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jessica Jeffrey, MD, MPH, MBA, Associate Professor of Psychiatry, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-000795
Record Dates: First submitted 2024-03-25; First posted 2024-04-09 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: PTSD, Post Traumatic Stress Disorder; Adolescents; Psychotherapy
Keywords: PTSD; MDMA; Adolescent; Psychotherapy
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- MDMA Psychotherapy (Experimental): Open-label fixed-dose trial whereby 10 youth with treatment-resistant PTSD will be recruited. Treatment-resistant depression is defined as having continued DSM-5 diagnosis of PTSD following at least 3 months of psychotherapy and (either separately or combined) at least 3 months SSRI pharmacotherapy. Prior to entering the trial, youth will undergo a preliminary medical and psychiatric screening to determine eligibility. Eligible youth will then proceed to 3-month MDMA-assisted psychotherapy, which includes 13 sessions of psychotherapy with two MDMA experimental medication sessions of 80mg and 120mg, respectively. Study assessments will include a baseline assessment, weekly assessments throughout the course of the treatment trial, and assessments at 3 months and 6 months post-treatment.
  Interventions: Drug: MDMA; Behavioral: Psychotherapy

INTERVENTIONS:
Drug: MDMA — MDMA will be dosed in pre-filled capsules and administered orally to participants in two fixed doses - an 80mg dose following the fourth session and a 120mg dose following the ninth session of MDMA to each participant. MDMA experimental medication administration session 1 (8 hours); MDMA experimental medication session 2 (8 hours). Participants will be required to remain in the therapy room for the duration of the experimental medication sessions without the youths' parent/guardian present. The parent/guardian will be invited to attend integration sessions and must be available to drop off and pick up the participant.
Behavioral: Psychotherapy — Treatment session order: Four weekly 90-minute experimental medication preparation psychotherapy sessions; four weekly 90-minute psychotherapy integration sessions, starting the day following the preceding experimental medication session; and Five weekly 90-minute psychotherapy integration sessions, starting the day following the preceding experimental medication session.

SUMMARY:
The primary objective of this study is to determine the safety and feasibility of 3,4-methylenedioxymethamphetamine (MDMA) -assisted psychotherapy to treat resistant post-traumatic stress disorder (PTSD). The secondary objectives are the exploration of effectiveness for treatment-resistant PTSD, symptoms of depression, and anxiety symptoms.

DETAILED DESCRIPTION:
This study is an open-label fixed dose trial whereby youth with treatment-resistant post-traumatic stress disorder (PTSD) will be recruited. Treatment-resistant depression is defined as having continued Diagnostic Statistical Manual (DSM-5) diagnosis of PTSD following at least 3 months of psychotherapy and (either separately or combined) at least 3 months of SSRI pharmacotherapy. Before entering the trial, youth will undergo a preliminary medical and psychiatric screening to determine eligibility. Eligible youth will then proceed to 3-month MDMA-assisted psychotherapy, which includes 13 sessions of psychotherapy with two MDMA experimental medication sessions of 80mg and 120mg, respectively. Study assessments will include a baseline assessment, weekly assessments throughout the course of the treatment trial, and assessments at 3 months and 6 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet DSM-5 criteria for current PTSD in response to a traumatic experience. An individual is not excluded if they experience more than one traumatic event. (Traumatic Event Screening Inventory for Children given to youth and caregiver, youth given CPSS if positive screen.)
* Participants must have treatment-resistant PTSD, as defined by having continued diagnosis of PTSD following at least 3-months of psychotherapy and pharmacotherapy. Psychotherapeutic treatments may include, but are not limited to, cognitive behavioral therapy (including trauma-focused cognitive behavioral therapy and exposure therapy, stress inoculation training, including anxiety management, and insight-oriented psychotherapy). Pharmacotherapies include selective serotonin reuptake inhibitors (SSRIs).
* Participants may also meet criteria for a mood (except bipolar disorder) or anxiety disorder. The inclusion of adolescents with either mood or anxiety disorders is essential given frequency of co-occurring disorders.
* Participants must be 16-17 years old at time of study screening.
* Participants; parents/caregivers must be willing to commit to two experimental sessions, therapy sessions, follow-up sessions, and completion of assessment parameters and instruments. Adolescents must assent.
* Participants must be willing to refrain from taking any psychotropic medication from the outset of the study until follow-up at 3 months. The scheduled outcome measures at 6 months will be conducted regardless of whether additional psychotropic medication was used. If they are being treated with psychoactive drugs at the time they are recruited into the study, agreement to suspend treatment must be obtained in writing from their outside treating physician. The drugs would be tapered in an appropriate fashion to avoid withdrawal effects (interval of at least five times the half-life).
* Participants who are in ongoing psychotherapy at the time they are recruited into the study may continue to see their outside therapist during the course of the study. If they desire that the investigators communicate directly with the therapist, parents/caregivers must sign a release of information. They may not change therapists, increase the length and frequency of sessions, or commence a new type of therapy until one month following the second experimental medication session.
* Participants must agree that, for one week preceding each experimental session: They will refrain from taking any herbal supplement (except with prior approval of the research team). They will not take any nonprescription medications (with the exception of NSAIDs or acetaminophen unless with prior approval of the research team). Without the permission of their physician, they will not take any prescription medications (with the exception of birth control pills, thyroid hormones or other medications approved by the research team).
* Participants must agree to take nothing my mouth except alcohol-free liquids after midnight the evening before the experimental sessions. Patient must also refrain from the use of psychoactive substances, including caffeine and cannabis, within 24 hours of the experimental sessions and for 24 hours following the experimental sessions.
* Participants must be willing to be driven home by their parent/caregiver the evening of the experimental sessions and return with their parent/caregiver the following morning for the first integration therapy sessions.
* Participants must be willing to be contacted via telephone on a daily basis by one of the investigators for a week after the experimental sessions.
* Participants who do not adhere to the usual progression of scheduled visits, as may occur when a session is delayed, must agree to maintain weekly telephone contact with the study investigators, and must agree to speak with the investigators if there is a significant increase in symptoms for which they were previously medicated, if there is unanticipated need to contact their treating therapist, or if there are any changes in medication.
* Female participants must have a negative pregnancy test at study intake and must agree to use of an effective form of birth control.
* Participants must have sufficient proficiency in English to participate in psychotherapy in English. They and their parents/caregivers must be fluent in English and able to understand documents in English.

Exclusion Criteria:

* Participants who are experiencing current or at imminent risk for trauma and victimization as assessed by information gathered during the screening.
* Participants who appear to reside within an unsupportive and/or chaotic family structure (ex: Department of Child and Family Services (DCFS) involvement).
* Sexually active females who are not practicing an effective means of birth control.
* Participants with a personal or first-degree family history of a primary psychotic disorder or bipolar affective disorder.
* Participants with a personal history of an eating disorder, dissociative identity disorders, or borderline personality disorder.
* Participants with evidence or history of significant hematological, endocrine, cerebrovascular, cardiovascular, coronary, pulmonary, renal, gastrointestinal, immunocompromising, or neurological disease, including seizure disorder. Participants with hypothyroidism who are stable on thyroid replacement will not be excluded.
* Any of the following cardiovascular conditions: hypertension, coronary artery disease, peripheral vascular disease, congenital long QT syndrome, cardiac hypertrophy, cardiac ischemia, congestive heart failure, tachycardia, artificial heart valve, or any other significant cardiovascular condition.
* Resting blood pressure above 140 systolic, 90 diastolic (averaged across four separate measurements)
* Participants with hepatic disease, or history of hyponatremia or hyperthermia.
* Participants weighing less than 50 kg (30th percentile for 16 years and 25th percentile for 17 years) or more than 105 kg.
* Participants reporting any prior use of "ecstasy", methamphetamine, cocaine, heroin, misuse of prescription opiates or benzodiazepines.
* Participants meeting DSM 5 criteria for a substance use disorder.
* Participants with previous history of psychiatric hospitalization.
* Participants who would present with significant current suicidality (as measured by PHQ-9 and CRRRS) or who are deemed by the study team to need a higher level of care than the outpatient treatment the study is providing.
* Participants requiring ongoing concomitant therapy with psychoactive drug and unwilling or unable to taper off the medication(s) under physician supervision.
* Any participant whose parent/caregiver is not able to give adequate informed consent or any participant who is not able to give assent.

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in heart rhythm via Carnation Ambulatory Heart Monitor | Throughout the 24 hours prior to each experimental medication session, throughout the duration of each drug administration session, and the 24 hours following each experimental medication session. Up to 64 hours.
  Changes in heart rhythm via Carnation Ambulatory Heart Monitor
Changes in blood pressure | Baseline assessment and at 1-hour intervals throughout each experimental medication session. Up to 17 hours total.
  changes in blood pressure as measured by blood pressure machine
Change in pulse | Baseline assessment and at 1-hour intervals throughout each experimental medication session. Up to 17 hours total.
  Change in pulse as part of measuring vitals
Change in body temperature | Baseline assessment and at 1-hour intervals throughout each experimental medication session. Up to 17 hours total
  Changes in body temperature as measured by thermometer
Mean change in score of visual analog scale to assess potential for misuse of MDMA | Weekly throughout treatment and at 3-month and 6-month follow-ups. Through study completion, an average of 9 months
  Investigate MDMA drug abuse potential through visual analog scale. Range for scale is 1-5 and will ask about the likability of the substance and the desire to use it in a non-clinical context.

SECONDARY OUTCOMES:
Mean change in PTSD symptom severity via the Child PTSD Symptom Scale | Baseline, One month Post Experimental Session, and 3 and 6 months post-treatment. Through study completion, an average of 9 months
  Change in PTSD symptom severity via the Child PTSD Symptom Scale (CPSS). The Child PTSD Symptom Scale (CPSS) measures posttraumatic stress disorder diagnosis and severity in the past month in children aged 8 to 18. Possible scores range from 0 to 80, with higher scores indicating a worse outcome/greater severity of symptoms.
Mean change in PTSD symptom severity via the Clinician-Administered PTSD Scale (CAPS-CA-5) | Baseline, One month Post Experimental Session, and 3 and 6 months post-treatment. Through study completion, an average of 9 months
  Change in PTSD symptom severity via the CAPS-CA-5. The Clinician-Administered PTSD Scale(CAPS-CA-5) measures posttraumatic stress disorder symptoms in the past month in children aged 7 and above. Possible scores range from 0 to 80 , with higher scores indicating more severe PTSD symptoms.
Mean change in depression symptom severity via the Patient Health Questionnaire-9 (PHQ-9). | Baseline and at each study visit following MDMA experimental medication sessions. Through study completion, an average of 9 months
  Change in depressive symptom severity via the PHQ-9. The Patient Health Questionnaire-9 (PHQ-9) measures the severity of depression. Possible scores range from 0 to 27, with higher scores indicating greater severity of depressive symptoms.
Mean change in anxiety symptom severity via the Generalized Anxiety Disorder 7-item (GAD-7) | Baseline and at each study visit following the experimental medication sessions. Through study completion, an average of 9 months
  Change in Anxiety symptoms assessed by the GAD-7. Generalized Anxiety Disorder 7-item scale measures the severity of anxiety. Possible scores range from 0 to 21, with higher scores indicating greater anxiety severity.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Semel Institute for Neuroscience and Human Behavior, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No